CLINICAL TRIAL: NCT00841295
Title: Effects of Parenteral L-carnitine Supplementation in Premature Neonates
Acronym: CarniPrema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PHRI06-FL / CARNIPREMA; N° EudraCT: 2007-002446-37 (Other: N° EudraCT); Réf.CPP: 2007-R24 (Other: CPP Tours); Réf.Afssaps: A70583-46 (Other: AFSSaPS)
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Complication of Prematurity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carnitine (Experimental): Intervention 'Parenteral L-carnitine supplementation' Parenteral carnitine supplementation (9 ± 1 mg/kg/d), from day 4, until than enteral nutrition provides sufficient carnitine source.
  Interventions: Drug: Parenteral L-carnitine supplementation
- Controle (Placebo Comparator): Intervention 'Parenteral supplementation with sterile water'
  Interventions: Drug: Parenteral supplementation with sterile water

INTERVENTIONS:
Drug: Parenteral L-carnitine supplementation — Parenteral carnitine supplementation (9 ± 1 mg/kg/d), from day 4, until than enteral nutrition provides sufficient carnitine source.
  Arms: Carnitine
Drug: Parenteral supplementation with sterile water — Parenteral supplementation with an equivalent volume of sterile water
  Arms: Controle

SUMMARY:
Background: Carnitine is the essential cofactor for various enzyme activities of human metabolism, especially for the mitochondrial carnitine shuttle that transfers long-chain fatty acids as acylcarnitine esters across the inner mitochondrial membrane for Beta-oxidation and energy production. Intracellular carnitine deficiency induces an impairment of long-chain fatty acid oxidation. In human, approximately 75% of carnitine comes from the diet and 25% from endogenous liver synthesis. In the neonatal period, more specifically in the premature, liver synthesis capacity is reduced because of immaturity of the biosynthetic pathway, and carnitine levels are related to exogenous sources. Traditionally, carnitine is not added to parenteral nutrition. Indeed, without enteral feeds and carnitine supplementation of parenteral nutrition, preterm infants' plasma carnitine levels fall during the first weeks of life, particularly in subjects requiring a prolonged exclusive parenteral nutrition. The potential deleterious role of carnitine deficiency has not been clearly demonstrated in these infants. However, most patients with primary carnitine deficiency, a genetic defect of carnitine transport inducing a severe carnitine deficiency, commonly develop liver symptoms (encompassing visceral steatosis, hyperammonemia and recurrent hypoketotic hypoglycemias) and/or cardiomyopathy and myopathy. In these latter patients, carnitine supplementation improves all the symptoms.

Hypothesis: Carnitine deficiency of the premature and very low birth weight infants may be one of the factors involved in the liver disease frequently associated with prolonged parenteral nutrition, and may have deleterious effects on cardiac and muscle metabolism and functions.

Aims: To demonstrate beneficial effects of parenteral carnitine supplementation in premature neonates for liver, heart and muscle metabolism and functions.

Study Type: Multicentric prospective and randomised study

Subjects: Premature and very low birth weight neonates, defined by gestational age minor or equal to 28 weeks and/or birth weight minor or equal to 1000 grams, 80 subjects will be enrolled during 2.5 years

Interventions: Arm 1 (experimental): parenteral carnitine supplementation (9 ± 1 mg/kg/d), from day 4, until than enteral nutrition provides sufficient carnitine source; Arm 2 (Placebo comparator): parenteral supplementation with an equivalent volume of sterile water.

DETAILED DESCRIPTION:
Background: Carnitine is the essential cofactor for various enzyme activities of human metabolism, especially for the mitochondrial carnitine shuttle that transfers long-chain fatty acids as acylcarnitine esters across the inner mitochondrial membrane for Beta-oxidation and energy production. Intracellular carnitine deficiency induces an impairment of long-chain fatty acid oxidation. In human, approximately 75% of carnitine comes from the diet and 25% from endogenous liver synthesis. In the neonatal period, more specifically in the premature, liver synthesis capacity is reduced because of immaturity of the biosynthetic pathway, and carnitine levels are related to exogenous sources. Traditionally, carnitine is not added to parenteral nutrition. Indeed, without enteral feeds and carnitine supplementation of parenteral nutrition, preterm infants' plasma carnitine levels fall during the first weeks of life, particularly in subjects requiring a prolonged exclusive parenteral nutrition. The potential deleterious role of carnitine deficiency has not been clearly demonstrated in these infants. However, most patients with primary carnitine deficiency, a genetic defect of carnitine transport inducing a severe carnitine deficiency, commonly develop liver symptoms (encompassing visceral steatosis, hyperammonemia and recurrent hypoketotic hypoglycemias) and/or cardiomyopathy and myopathy. In these latter patients, carnitine supplementation improves all the symptoms.

Hypothesis: Carnitine deficiency of the premature and very low birth weight infants may be one of the factors involved in the liver disease frequently associated with prolonged parenteral nutrition, and may have deleterious effects on cardiac and muscle metabolism and functions.

Aims: To demonstrate beneficial effects of parenteral carnitine supplementation in premature neonates for liver, heart and muscle metabolism and functions.

Study Type: Multicentric prospective and randomised study

Subjects: Premature and very low birth weight neonates, defined by gestational age minor or equal to 28 weeks and/or birth weight minor or equal to 1000 grams, 80 subjects will be enrolled during 2.5 years

Interventions: Arm 1 (experimental): parenteral carnitine supplementation (9 ± 1 mg/kg/d), from day 4, until than enteral nutrition provides sufficient carnitine source; Arm 2 (Placebo comparator): parenteral supplementation with an equivalent volume of sterile water.

Primary Outcome: Plasma Gamma Glutamyl Transferase level after 21 days of parenteral supplementation.

Secondary Outcomes: Short- (during parenteral supplementation) and long- (3 to 5 months of age) term outcomes: 1) Liver function (levels of ammonemia, hyaluronic acid, bilirubin, prothrombin time test, ursodeoxycholic acid therapy), 2) cardiac function (echocardiography, EKG), 3) muscle integrity (CK levels), 4) neurological injuries (brain ultrasound and MRI), 5) respiratory immaturity, 6) acylcarnitine profile and other fatty acid derivatives.

Expected Findings: Systematic parenteral carnitine supplementation will prevent systemic carnitine deficiency, and will improve liver dysfunction (decreased duration and severity of liver disease) associated with prolonged parenteral nutrition, will improve cardiac and muscle functions, and will prevent cerebral injury in premature infants with very low birth weight.

ELIGIBILITY:
Inclusion Criteria:

* Premature newborn admitted in Intensive Care Unit,
* Gestational age minor or equal than 28 weeks and 6 days,
* Needing prolonged parenteral nutrition through a central intravenous catheter,
* Parenteral nutrition started before 6 days of life,
* Both parents (or legal tutor) gave written informed consent for their children,
* Patient affiliated to "Sécurité Sociale" of his parents.

Exclusion Criteria:

* Severe associated disorder, with a probable short-term death,
* Identified genetic disease,
* Polymalformative syndrome, or severe malformation (heart, brain, others…),
* Inborn error of metabolism,
* Probable transfer of the subject before 25 days of life in another hospital that do not collaborate to this study.

Max Age: 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2008-07; Primary Completion 2013-03 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Plasma Gamma Glutamyl Transferase level | After 21 days of parenteral supplementation.

SECONDARY OUTCOMES:
Liver function: levels of ammonemia, hyaluronic acid, bilirubin, prothrombin time test, use of ursodeoxycholic acid therapy. | Short- (during parenteral supplementation) and long- (3 to 5 months of age) term outcome
Cardiac function: echocardiography, EKG. | Short- (during parenteral supplementation) and long- (3 to 5 months of age) term outcome
Muscle integrity: CK levels. | Short- (during parenteral supplementation) and long- (3 to 5 months of age) term outcome
Neurological injuries: brain ultrasound and MRI. | Short- (during parenteral supplementation, ultrasound) and long- (3 to 5 months of age, MRI) term outcome
Respiratory immaturity | Short- (during parenteral supplementation) and long- (3 to 5 months of age) term outcome
Acylcarnitine profile, and other fatty acid derivative levels. | Short- (during parenteral supplementation) and long- (3 to 5 months of age) term outcome

CONTACTS AND LOCATIONS:
Overall Officials: François LABARTHE, MD, Principal Investigator — University Hospital, Tours
Locations (2):
- France (2):
  - UH Porte Madeleine, Orléans
  - Hôpital Clocheville, University Hospital, Tours, Tours